CLINICAL TRIAL: NCT06590844
Title: Exploratory Study on the Efficacy and Safety of "cindilizumab + Bevacizumab + Coenzyme I for Injection" in Unresectable Hepatocellular Carcinoma
Brief Title: "cindilizumab + Bevacizumab + Coenzyme I for Injection" in Unresectable Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNPD1
Record Dates: First submitted 2024-03-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental group (Experimental): On the first day, we will treat patients with Tybo Sulsintilimab ® 200mg IV and Dalutin ® Bevacizumab 15mg/kg IV every 21 days. The first to third days were treated with injectable coenzyme I, 100mg/day IV, every 21 days as a cycle.
  Interventions: Drug: Injectable coenzyme I

INTERVENTIONS:
Drug: Injectable coenzyme I — On the first day, we will treat patients with Tybo Sulsintilimab ® 200mg IV and Dalutin ® Bevacizumab 15mg/kg IV every 21 days. The first to third days were treated with injectable coenzyme I, 100mg/day IV, every 21 days as a cycle.

SUMMARY:
This study is a single-arm, single-center, non-randomized, open-label study. A total of 37 patients with locally advanced or metastatic HCC who have not received systemic therapy, are not suitable for radical surgical resection or local treatment, or have disease progression after surgical resection or local treatment, the efficacy and safety of "cindilizumab + bevacizumab + coenzyme I for injection" are initially explored.

DETAILED DESCRIPTION:
1. Background According to the latest global cancer burden data for 2020 released by the World Health Organization Agency for International Research on Cancer (IARC), about 390,000 people die from liver cancer every year, accounting for 47 percent of the global liver cancer deaths. As the second mortality malignant tumor in China, the five-year survival rate is only 14%. Based on the ORIENT-32 study, the first PD-1 immunosuppressive combination therapy sindilizumab combined with bevacizumab for the first-line treatment of patients with advanced liver cancer has been officially approved by the National Drug Administration for the first-line treatment of unresectable or metastatic liver cancer."Sindilizumab + bevacizumab" marks a breakthrough in liver cancer immunotherapy with the combination of PD-1 immunosuppressive agents. However, clinical trial data showed that the response rate of immunosuppressive agents in solid tumors was low (ORIENT-32 ORR of "Sindilizumab + bevacizumab" regimen was 25%) and susceptible to tolerance. Therefore, finding effective efficacy predictive markers and combination therapy is an important method to improve the effect of tumor immunotherapy and promote tumor precision immunotherapy.

Coenzyme I (nicotinamide adenine dinucleotide, NAD+) Is a very important coenzyme in biological redox reactions and plays a crucial role in various biological processes including metabolism, senescence, cell death, DNA repair and gene expression。NAD+Metabolic abnormalities are closely related to the occurrence and development of many diseases, including cancer. On November 9,2020, Academician Wang Hongyang's team published the title "NAD" on Cell Metabolism+metabolism maintains inducible PD-L1 expression to drive tumor immune evasion " research paper, reveals the NAD+Metabolism drives novel mechanisms of tumor immune escape by regulating immune checkpoint PD-L1 expression, and is proposed by supplementing NAD+Novel strategies to enhance therapeutic sensitivity of anti-PD-1 / PD-L1 antibodies[5]. Further studies found that the anti-PD-1 antibody suppressed tumor burden by 42.2% in a model of Hep 1-6-CD38 immunotherapy administered NAD+The tumor burden suppression rate after the combination therapy was 82.8%. In the primary tolerance model of Pan02 immunotherapy in pancreatic cancer, the anti-PD-1 antibody suppressed tumor burden by only 18.6%, giving NAD+The combined treatment tumor burden suppression rate was 64.7%. In both models simultaneously, the NAD+The group alone did not promote tumor growth compared with the control group. The study has important clinical implications to complement the NAD+A combination regimen with anti-PD-1 / PD-L1 antibodies could provide a novel therapeutic strategy for tumors resistant to immunotherapy.

2、Effectiveness evaluation indicators (primary efficacy indicators and secondary efficacy indicators) Primary endpoint

* ORR as assessed by mRECIST 1.1 Selected secondary study endpoints and exploratory endpoints
* Safety and tolerability
* DOR, DCR, PFS, TTP, OS, as assessed by mRECIST 1.1
* Conversion rate Safety evaluation index The incidence and severity of all adverse events (AEs), treatment emergent adverse events (TEAEs), grade 3 or higher study drug-related adverse events, serious adverse events (SAEs) were judged according to CTCAE V5.0, and the clinical characteristics, severity, time of occurrence of any adverse events were recorded, End time, duration, treatment measures, and outcomes, and determine their relevance to treatment regimens.

  3、Statistical Methods All statistical analyses will be performed in SAS 9.4 or later. In general, continuous variables will be statistically described using the number of cases, mean, median, standard deviation, minimum and maximum values; Categorical and hierarchical variables will be statistically described using the frequency and percentage of each category or grade, and missing values will not be included in the calculation of percentages unless otherwise indicated. Unless otherwise stated, all statistical tests will be performed using a two-sided test of α = 0.05 with a two-sided 95% confidence interval (CI) calculated.

  4、Statistical processing All statistical analyses will be performed using SAS 9.4 or later. In general, continuous variables will be statistically described using the number of cases, mean, median, standard deviation, minimum and maximum values; Categorical and hierarchical variables will be statistically described using the frequency and percentage of each category or grade, and missing values will not be included in the calculation of percentages unless otherwise indicated. Unless otherwise stated, all statistical tests will be performed using a two-sided test of α = 0.05 with a two-sided 95% confidence interval (CI) calculated.

  5、Data security monitoring The clinical study will develop a data security monitoring plan according to the size of the risk. All adverse events are recorded in detail, properly handled and tracked until properly resolved or the condition is stable, and serious adverse events and unexpected events are reported to the ethics committee, competent authorities and drug regulatory departments in a timely manner in accordance with regulations; The principal investigator conducted a systematic review of all adverse events on a regular basis, and convened investigator meetings to assess the risks and benefits of the study if necessary; Double-blind trials can be urgently unblinded if necessary to ensure the safety and rights of subjects; For studies with greater than minimal risk, an independent data monitor will be assigned to monitor the study data, and for high-risk studies, an independent data safety monitoring committee will be established to monitor the accumulated safety data and efficacy data to make recommendations on whether to proceed with the study.

  6、Ethics of clinical research Clinical studies will follow the Declaration of Helsinki and other relevant regulations of the World Medical Assembly. The study can only be carried out after the approval of the study by the ethics committee before the start of the study. Before each subject is enrolled in this study, the investigator has the responsibility to fully and comprehensively introduce the purpose, procedures and possible risks of this study to the subject or his agent, and sign a written informed consent form, and the subject should be let know that they have the right to withdraw from this study at any time, and the informed consent should be retained as a clinical study document for future reference. The privacy and confidentiality of the subjects will be protected during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytologically confirmed hepatocellular carcinoma, or cirrhosis of the liver meets the American Association for the Study of Liver Diseases (AASLD) clinical diagnostic criteria for hepatocellular carcinoma.
2. 18 years old≤ age ≤ 80 years old
3. ECOG PS 0-1 points, Child-Pugh score ≤7 points.
4. The 2022 edition of the Guidelines for the Diagnosis and Treatment of Liver Cancer of the National Health Commission of China is stage IIb and above.
5. Have not received systemic anti-tumor therapy for HCC before the first dose (enrollment is allowed more than 6 months after the end of postoperative adjuvant chemotherapy), and enrollment is allowed 28 days after the end of TACE treatment.
6. Have adequate organ and bone marrow function. The laboratory test values within 7 days prior to enrollment meet the following requirements:

   1. Routine blood count: absolute neutrophil count (ANC) ≥1.5× 109/L; Platelet count (PLT) ≥ 75×10 9/L; Hemoglobin content (HGB) ≥ 9.0 g/dL.
   2. Liver function: serum total bilirubin (TBIL) ≤2× upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5×ULN; serum albumin≥ 28 g/L; Alkaline phosphatase (ALP) ≤5×ULN.
   3. Renal function: serum creatinine (Cr) ≤ 1.5× ULN or creatinine clearance (CCr) ≥ 50mL/min; Patients with a urine protein ≥ 2+ should have a 24-hour urine collection and a 24-hour urine protein quantification <1 g.
   4. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN.
7. Patients with acute or chronic active hepatitis B or hepatitis C infection, hepatitis B virus (HBV) DNA less than 2000IU/ml or 10 copies/ml; Hepatitis C virus (HCV) RNA is less than 1000 copies/ml.

Agree to participate in this clinical trial and sign a written informed consent form..

Exclusion Criteria:

1. Previously confirmed fibrolamellarhepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma and other components previously confirmed by histology/cytology.
2. Have a history of hepatic encephalopathy, or have a history of liver transplantation.
3. The portal vein trunk cancer thrombus involves the contralateral portal vein branch at the same time, or the superior mesenteric vein and inferior vena cava cancer thrombus at the same time..
4. Pleural effusion, ascites, and pericardial effusion that need to be drained with clinical symptoms.
5. Hepatitis B surface antigen (HbsAg) is positive at the same time as anti-HCV antibodies.
6. There are central nervous system metastases.
7. HIV infection.
8. Gastroscopy showed positive red sign of esophageal and gastric varices.
9. Women who are pregnant or preparing to become pregnant or breastfeeding.
10. Those who are known to be allergic to coenzyme I and its components or have serious adverse reactions.
11. Those who have participated in other clinical trials within 3 months before participating in this trial.
12. In the judgment of the investigator, the patient is unable to complete this study or is unable to comply with the requirements of this study.
13. Participating in other interventional clinical trials.

Ages: 18 Days to 80 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
ORR | 4-6 weeks
  ORR as assessed by mRECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Liangxin Liu, Professor, Principal Investigator — AnhuiI Provincial Hospital
Locations (1):
- AnhuiI Provincial Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No